CLINICAL TRIAL: NCT00567424
Title: An Open-label Evaluation of Drug Interactions, Safety, Tolerability and Efficacy of GW273225 Add-on Treatment of Partial Seizures, Whether or Not Secondarily Generalized
Brief Title: GW273225 Therapy Added To Current Seizure Treatments In Patients With Partial Seizures
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No longer viable
Sponsor: GlaxoSmithKline (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEC107055
Record Dates: First submitted 2006-07-20; First posted 2007-12-05 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Epilepsy
Keywords: epilepsy; refractory; seizure; drug interactions; pharmacokinetics
MeSH Terms: conditions — Epilepsy; Seizures

INTERVENTIONS:
Drug: GW273225

SUMMARY:
Study to determine drug interactions between GW273225 and the anticonvulsants valproate, carbamazepine or phenytoin

ELIGIBILITY:
Inclusion criteria:

* Confident diagnosis of epilepsy
* Currently on VPA, CBZ or PHT
* >or= 4 seizures/4 weeks prior to screen

Exclusion criteria:

* Prior lamotrigine use (excluded if treatment discontinued for clinically significant safety reasons (i.e., rash, hypersensitivity)).
* Females of childbearing potential on hormonal contraceptives or hormone replacement therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-07; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic drug interactions with the most common inhibiting and inducing antiepileptic drugs AEDs: valproate(VPA), carbamazepine(CBZ) and phenytoin (PHT).

SECONDARY OUTCOMES:
Safety/tolerability of GW273225 in adults with refractory epilepsy Efficacy of GW273225 in adults with refractory epilepsy Potential initial starting doses for a subsequent placebo-controlled dose-ranging Phase IIb study.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (29):
- United States (29):
  - GSK Clinical Trials Call Center, Phoenix, Arizona
  - GSK Clinical Trials Call Center, Sun City, Arizona
  - GSK Clinical Trials Call Center, Little Rock, Arkansas
  - GSK Clinical Trials Call Center, San Jose, California
  - GSK Clinical Trials Call Center, Santa Monica, California
  - GSK Clinical Trials Call Center, Jacksonville, Florida
  - GSK Clinical Trials Call Center, Tallahassee, Florida
  - GSK Clinical Trials Call Center, Tampa, Florida
  - GSK Clinical Trials Call Center, Chicago, Illinois
  - GSK Clinical Trials Call Center, Springfield, Illinois
  - GSK Clinical Trials Call Center, Iowa City, Iowa
  - GSK Clinical Trials Call Center, Wichita, Kansas
  - GSK Clinical Trials Call Center, Baltimore, Maryland
  - GSK Clinical Trials Call Center, Boston, Massachusetts
  - GSK Clinical Trials Call Center, Rochester, Minnesota
  - GSK Clinical Trials Call Center, Saint Cloud, Minnesota
  - GSK Clinical Trials Call Center, Springfield, Missouri
  - GSK Clinical Trials Call Center, St Louis, Missouri
  - GSK Clinical Trials Call Center, Amherst, New York
  - GSK Clinical Trials Call Center, Durham, North Carolina
  - GSK Clinical Trials Call Center, Cleveland, Ohio
  - GSK Clinical Trials Call Center, Toledo, Ohio
  - GSK Clinical Trials Call Center, Medford, Oregon
  - GSK Clinical Trials Call Center, Portland, Oregon
  - GSK Clinical Trials Call Center, Dallas, Texas
  - GSK Clinical Trials Call Center, Burlington, Vermont
  - GSK Clinical Trials Call Center, Richmond, Virginia
  - GSK Clinical Trials Call Center, Roanoke, Virginia
  - GSK Clinical Trials Call Center, Seattle, Washington